CLINICAL TRIAL: NCT06428396
Title: A Phase 2, Randomized, Active-controlled, Open-label, Multicenter Study of Belzutifan Plus Fulvestrant in Participants With Estrogen Receptor Positive, HER2 Negative Unresectable Locally Advanced or Metastic Breast Cancer After Progression on Previous Endocrine Therapy (LITESPARK-029)
Brief Title: Study of Belzutifan (MK-6482) Plus Fulvestrant for ER+/HER2- Metastatic Breast Cancer (MK-6482-029/LITESPARK-029)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6482-029; MK-6482-029 (Other: MSD); LITESPARK-029 (Other: MSD)
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — belzutifan; Fulvestrant; Everolimus; exemestane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Belzutifan + Fulvestrant (Experimental): Participants will receive belzutifan 120 mg orally once daily (QD) PLUS fulvestrant 500 mg via intramuscular (IM) injection on Days 1 and 15 of Cycle 1, and Day 1 of each 28-day cycle thereafter until progressive disease or discontinuation.
  Interventions: Drug: Belzutifan; Drug: Fulvestrant
- Everolimus + ET (fulvestrant or exemestane) (Active Comparator): Participants will receive everolimus 10 mg orally QD PLUS investigator's choice of fulvestrant 500 mg via IM injection on Days 1 and 15 of Cycle 1, and Day 1 of each 28-day cycle thereafter OR exemestane 25 mg orally QD until progressive disease or discontinuation.
  Interventions: Drug: Fulvestrant; Drug: Everolimus; Drug: Exemestane

INTERVENTIONS:
Drug: Belzutifan — Belzutifan 120 mg administered QD as an oral tablet.
  Other Names: MK-6482
  Arms: Belzutifan + Fulvestrant
Drug: Fulvestrant — Fulvestrant 500 mg administered as an IM injection.
Drug: Everolimus — Administered at 10mg via oral tablets QD.
  Arms: Everolimus + ET (fulvestrant or exemestane)
Drug: Exemestane — Administered at 25 mg via oral tablets QD.
  Arms: Everolimus + ET (fulvestrant or exemestane)

SUMMARY:
The purpose of this study is to assess the efficacy and safety of belzutifan (MK-6482) plus fulvestrant compared to everolimus plus endocrine therapy (ET) (investigator's choice of fulvestrant or exemestane) in adults with estrogen receptor-positive, human epidermal growth factor receptor 2-negative (ER+/HER2-) unresectable metastatic breast cancer. There is no formal hypothesis testing in this study.

ELIGIBILITY:
Inclusion Criteria:

* Has a diagnosis of estrogen receptor positive (ER+)/human epidermal growth factor receptor negative (HER2-) invasive breast carcinoma that is either locally advanced disease not amenable to resection or metastatic disease not treatable with curative intent
* Has documented radiographic confirmation of disease progression during or after the last administered endocrine therapy (ET)
* Provides additional tissue from the same sample used to determine ER and HER2 status locally
* Has received ET in the noncurative setting and has 1) Radiographic disease progression on 12 months or more of ET in combination with CDK4/6 inhibitor in the noncurative setting or 2) Received at least 2 lines of ET in the noncurative setting including CDK4/6 inhibitor where the CDK 4/6 inhibitor was discontinued due to intolerance
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of randomization
* Participants who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or baseline. Participants with endocrine-related AEs who are adequately treated with hormone replacement or participants who have ≤Grade 2 neuropathy are eligible
* Participants who are hepatitis B surface antigen (HBsAg) positive are eligible if they have received hepatitis B virus (HBV) antiviral therapy for at least 4 weeks prior to the first dose of study intervention and have undetectable HBV viral load prior to randomization

Exclusion Criteria:

* Has Breast cancer amenable to treatment with curative intent
* Is unable to receive any of the endocrine therapies (ETs) (ie, fulvestrant or exemestane)
* Has known difficulty in tolerating oral medications, unable to swallow orally administered medication, or conditions which would impair absorption of oral medications such as uncontrolled nausea or vomiting (ie, CTCAE =Grade 3 despite antiemetic therapy), ongoing gastrointestinal obstruction, motility disorder, malabsorption syndrome, or prior gastric bypass
* Has advanced/metastatic, symptomatic visceral spread at risk of rapidly evolving into life-threatening complications
* Has active, bleeding diathesis, or on oral anti-vitamin K medication
* Has history of noninfectious pneumonitis/interstitial lung disease including radiation pneumonitis that required steroids or has current pneumonitis/interstitial lung disease
* Has a known germline BRCA mutation (deleterious or suspected deleterious) and has received previous treatment with poly-ADP ribose polymerase (PARP) inhibition either in the adjuvant or metastatic setting
* Has received prior fulvestrant in the adjuvant, unresectable locally advanced, or metastatic setting
* Has received any line of cytotoxic chemotherapy or PARP inhibitor in the unresectable or noncurative advanced/metastatic setting
* Has received prior radiotherapy for non-central nervous system (CNS) disease or required corticosteroids for radiation-related toxicities including radiation pneumonitis, within 14 days of the first dose of study intervention
* Is currently receiving either a strong inhibitor or inducer of CYP3A4 that cannot be discontinued for the duration of the study
* Has received prior systemic anticancer therapy including investigational agents within 4 weeks before randomization
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has concurrent active Hepatitis B and Hepatitis C virus infection
* Has clinically significant cardiac disease, including unstable angina, acute myocardial infarction within 6 months from Day 1 of study medication administration, or New York Heart Association Class III or Class IV congestive heart failure
* Has not adequately recovered from major surgery or have ongoing surgical complications

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-27 (Actual); Primary Completion 2027-05-05 (Estimated); Study Completion 2028-10-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | Up to approximately 29 months
  PFS is defined as the time from randomization to the first documented disease progression per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) based on blinded independent central review (BICR) or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Progression-free Survival (PFS) at 6 months | Up to approximately 29 months
  PFS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the PFS rate at 6 months using the entire PFS data up to the cut-off date. The cut-off date is event-driven and estimated to be approximately 28 months.
Progression-free Survival (PFS) at 12 months | Up to approximately 29 months
  PFS data will be cumulated to a certain cut-off date and the analysis will be performed via Kaplan-Meier approach to estimate the PFS rate at 12 months using the entire PFS data up to the cut-off date. The cut-off date is event-driven and estimated to be approximately 28 months.
Overall Survival (OS) | Up to approximately 29 months
  OS is defined as the time from randomization to death due to any cause.
Objective Response Rate (ORR) | Up to approximately 29 months
  ORR is defined as the percentage of participants who have achieved confirmed Complete Response (CR: disappearance of all target lesions) or a Partial Response (PR: at least a 30% decrease in the sum of diameters of target lesions) per RECIST 1.1 as assessed by BICR.
Clinical Benefit Rate (CBR) | Up to approximately 29 months
  CBR is defined as the percentage of participants who have CR: Disappearance of all target lesions, PR: At least a 30% decrease in the sum of diameters of target lesions, or stable disease (SD: Neither sufficient decrease to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study) for ≥24 weeks per RECIST 1.1 as assessed by BICR.
Number of Participants Who Experience an Adverse Event (AE) | Up to approximately 46 months
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.
Number of Participants Who Discontinue Study Treatment Due To an AE | Up to approximately 46 months
  An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (41):
- United States (14):
  - City of Hope - Phoenix ( Site 0006), Goodyear, Arizona
  - Cedars Sinai Medical Center ( Site 0012), Beverly Hills, California
  - Moores Cancer Center at UC San Diego Health ( Site 0025), La Jolla, California
  - USC/Norris Comprehensive Cancer Center ( Site 0013), Los Angeles, California
  - USC Norris Oncology Hematology Newport Beach ( Site 0029), Newport Beach, California
  - Northwest Georgia Oncology Centers, a Service of Wellstar Cobb Hospital ( Site 0011), Marietta, Georgia
  - Southeastern Regional Medical Center ( Site 0010), Newnan, Georgia
  - CHRISTUS Highland ( Site 0005), Shreveport, Louisiana
  - Renown Regional Medical Center ( Site 0018), Reno, Nevada
  - MD Anderson Cancer Center at Cooper ( Site 0024), Camden, New Jersey
  - MD Anderson ( Site 0015), Houston, Texas
  - Mays Cancer Center ( Site 0022), San Antonio, Texas
  - SSM Health Dean Medical Group - South Madison Campus Health Research/Circuit Clinical ( Site 0034), Madison, Wisconsin
  - Medical College of Wisconsin - Froedtert Hospital ( Site 0014), Milwaukee, Wisconsin
- Argentina (7):
  - Centro de Investigaciones Metabólicas (CINME)-Oncology ( Site 0504), CABA, Buenos Aires
  - Hospital Británico de Buenos Aires-Oncology ( Site 0500), Ciudad Autónoma de Buenos Aires, Buenos Aires
  - Instituto de Investigaciones Clínicas Mar del Plata ( Site 0502), Mar del Plata, Buenos Aires
  - Instituto Alexander Fleming-Alexander Fleming ( Site 0505), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Allende - Cerro-Oncology ( Site 0506), Córdoba, Córdoba Province
  - Instituto de Oncología de Rosario ( Site 0501), Rosario, Santa Fe Province
  - Hospital Italiano de Córdoba ( Site 0508), Córdoba
- Jewish General Hospital ( Site 0400), Montreal, Quebec, Canada
- Chile (4):
  - Centro de Investigación del Maule ( Site 4106), Talca, Maule Region
  - FALP ( Site 4102), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 4108), Santiago, Region M. de Santiago
  - Bradfordhill ( Site 4100), Santiago, Region M. de Santiago
- Colombia (3):
  - IMAT S.A.S ( Site 1205), Montería, Departamento de Córdoba
  - Oncologos Del Occidente ( Site 1200), Pereira, Risaralda Department
  - Fundacion Valle del Lili ( Site 1204), Cali, Valle del Cauca Department
- South Korea (2):
  - Seoul National University Hospital ( Site 3100), Seoul
  - Samsung Medical Center ( Site 3101), Seoul
- Taiwan (3):
  - National Cheng Kung University Hospital ( Site 3300), Tainan
  - National Taiwan University Hospital ( Site 3301), Taipei
  - National Taiwan University Cancer Center ( Site 3302), Taipei
- Thailand (3):
  - Faculty of Medicine Siriraj Hospital ( Site 3500), Bangkoknoi, Bangkok
  - Faculty of Medicine - Khon Kaen University ( Site 3502), Muang, Changwat Khon Kaen
  - Songklanagarind Hospital ( Site 3501), Hat Yai, Changwat Songkhla
- United Kingdom (4):
  - The Royal Cornwall Hospital ( Site 1904), Truro, England
  - St Bartholomews Hospital ( Site 1900), London, London, City of
  - The Christie Hospital NHS Foundation Trust ( Site 1902), Withington, Manchester
  - Ipswich Hospital ( Site 1911), Ipswich, Suffolk

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/